CLINICAL TRIAL: NCT00492648
Title: An Extension Study to Evaluate the Persistence of the Immune Responses Induced by GSK Biologicals Zoster Vaccine, GSK324332A, Administered in Healthy Adult Subjects Aged 18-30 Years and 50-70 Years
Brief Title: Month 30 & 42 Extension Studies of CRD-004 Primary Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109671; 109674
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Herpes Zoster
Keywords: GSK Biologicals; Varicella Zoster Virus (VZV); Intracellular cytokine staining (ICS); Vaccine; Cell mediated immunity (CMI); Herpes Zoster (HZ); Shingles
MeSH Terms: conditions — Herpes Zoster; Chickenpox | interventions — Blood Specimen Collection

ARMS (2):
- GSK1437173A 18-30 Years Old Group (Experimental): Subjects aged 18 to 30 years old receiving 2 doses GSK1437173A vaccine in the primary study.
  Interventions: Procedure: Blood sampling for assay of persistence of immunogenicity
- GSK1437173A 50-70 Years Old Group (Experimental): Subjects aged 50 to 70 years old receiving 2 doses GSK1437173A vaccine in the primary study.
  Interventions: Procedure: Blood sampling for assay of persistence of immunogenicity

INTERVENTIONS:
Procedure: Blood sampling for assay of persistence of immunogenicity — Two blood samples: 30 and 42 months after first vaccination

SUMMARY:
The safety and immunogenicity of the GSK324332A vaccine has been evaluated up to Month 12 post-vaccination in the primary study. In the extension studies presented here, the persistence of the cellular and humoral immune responses will be evaluated 30 and 42 months after the first vaccination in young and elderly adults who received the GSK324332A vaccine. This protocol posting deals only with objectives & outcome measures of the extension phase at Months 30 and 42. No new recruitment will be done in these extension phases of the primary study. No vaccines are administered in this phase of the study.

DETAILED DESCRIPTION:
All subjects in these extension phases of the study were previously vaccinated with the investigational herpes zoster vaccine GSK1437173A. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

Further details on the primary study can be found on our GSK study register (https://www.gsk-studyregister.com/advanced-search) by searching on the GSK study identifier 101501.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study;
* Subjects who successfully completed the primary study and who did not receive Varilrix in the primary study;
* Written informed consent obtained from the subject;
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) within 1 month preceding the study start, or planned use during the study period;
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within three months prior to the first study procedure, including corticosteroids, except inhaled and topical steroids are allowed;
* Administration or planned administration of a vaccine not foreseen by the study protocol within 2 weeks before the first study procedure, with the exception of the Influenza vaccine, which can be administered 1 week preceding the first study procedure;
* Previous vaccination against HZ, except the study vaccine administered in the primary study;
* History of HZ (shingles);
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination;
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first study procedure or planned administration during the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-06-25 (Actual); Primary Completion 2008-06-23 (Actual); Study Completion 2008-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

REFERENCES:
- [Derived] Keersmaekers N, Ogunjimi B, Van Damme P, Beutels P, Hens N. An ODE-based mixed modelling approach for B- and T-cell dynamics induced by Varicella-Zoster Virus vaccines in adults shows higher T-cell proliferation with Shingrix than with Varilrix. Vaccine. 2019 May 1;37(19):2537-2553. doi: 10.1016/j.vaccine.2019.03.075. Epub 2019 Apr 8. PMID 30975567
- [Derived] Leroux-Roels I, Leroux-Roels G, Clement F, Vandepapeliere P, Vassilev V, Ledent E, Heineman TC. A phase 1/2 clinical trial evaluating safety and immunogenicity of a varicella zoster glycoprotein e subunit vaccine candidate in young and older adults. J Infect Dis. 2012 Oct;206(8):1280-90. doi: 10.1093/infdis/jis497. Epub 2012 Aug 7. PMID 22872734

RESULTS

PARTICIPANT FLOW:
Groups:
- GSK1437173A 18-30 Years Old Group: Subjects aged 18 to 30 years old primed with 2 doses GSK1437173A vaccine.
- GSK1437173A 50-70 Years Old Group: Subjects aged 50 to 70 years old primed with 2 doses GSK1437173A vaccine.
Period: Month 30 (109671 Study)
Arm/Group | GSK1437173A 18-30 Years Old Group | GSK1437173A 50-70 Years Old Group
Started | 4 | 30
Completed | 4 | 29
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Month 42 (109674 Study)
Arm/Group | GSK1437173A 18-30 Years Old Group | GSK1437173A 50-70 Years Old Group
Started | 3 | 20
Completed | 3 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1437173A 18-30 Years Old Group | GSK1437173A 50-70 Years Old Group | Total
Number analyzed (Participants) | 4 | 30 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: For Month 30 (109671 Study)
  Years | 22.3 (3.20) | 54.9 (4.19) | 51.6 (11.40)
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: For Month 42 (109674 Study)
  Years
    number analyzed (Participants) | 3 | 20 | 23
    (all) | 22.7 (3.79) | 56.0 (4.59) | 51.6 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: For Month 30 (109671 Study)
  Participants
    Female | 4 | 23 | 27
    Male | 0 | 7 | 7
Sex: Female, Male [Count of Participants; unit: Participants] — Population: For Month 42 (109674 Study)
  Participants
    number analyzed (Participants) | 3 | 20 | 23
    Female | 3 | 16 | 19
    Male | 0 | 4 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Frequencies of Glycoprotein E (gE)-Specific Cluster of Differentiation 4 (CD4) / CD8 T Cells With at Least Two Antigen-specific Cytokines: Interferon Gamma (IFN-γ), Interleukin 2 (IL-2), Tumor Necrosis Factor Alpha (TNF-α), CD 40 Ligand (CD40L).
Description: The analysis focused on those gE-specific CD4 T cells secreting at least two different cytokines among IFN-γ, IL-2, TNF-α, and CD40L as determined by intracellular cytokine staining (ICS). No analysis of the immunogenicity data on CD8 T cell response to gE was performed, since no long-term vaccine effect on gE-specific CD8 T cell response was detected.
Time Frame: At Month 30 after the first vaccination.
Population: The analysis was based on the According-to-Protocol (ATP) cohort for persistence, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available for the assay and time point assessed.
Measure: Mean (Standard Deviation); unit: gE-specific CD4 cells/million CD4 cells
Arm/Group | GSK1437173A 18-30 Years Old Group | GSK1437173A 50-70 Years Old Group
Number analyzed (Participants) | 4 | 29
gE-specific CD4 cells/million CD4 cells | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4). | 1184.7 (925.8)

2. Primary Outcome: Frequencies of Varicella Zoster Virus (VZV)-Specific CD4 / CD8 T Cells With at Least Two Antigen-specific Cytokines (IFN-γ, IL-2, TNF-α, CD40L).
Description: The analysis focused on those VZV-specific CD4 T cells secreting at least two different cytokines among IFN-γ, IL-2, TNF-α, CD40L as determined by intracellular cytokine staining (ICS). No analysis of the immunogenicity data on CD8 T cell response to VZV was performed, since no long-term vaccine effect on VZV-specific CD8 T cell response was detected.
Time Frame: At Month 30 after the first vaccination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: VZV-specific CD4 cells/million CD4 cells
Arm/Group | GSK1437173A 18-30 Years Old Group | GSK1437173A 50-70 Years Old Group
Number analyzed (Participants) | 4 | 29
VZV-specific CD4 cells/million CD4 cells | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4). | 707.4 (533.1)

3. Primary Outcome: Frequencies of Glycoprotein E (gE)-Specific CD4 / CD8 T Cells With at Least Two Antigen-specific Cytokines (IFN-γ, IL-2, TNF-α, CD40L).
Description: The analysis focused on those gE-specific CD4 T cells secreting at least two different cytokines among IFN-γ, IL-2, TNF-α, CD40L as determined by intracellular cytokine staining (ICS). No analysis of the immunogenicity data on CD8 T cell response to gE was performed, since no long-term vaccine effect on gE-specific CD8 T cell response was detected.
Time Frame: At Month 42 after the first vaccination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gE-specific CD4 cells/million CD4 cells
Arm/Group | GSK1437173A 18-30 Years Old Group | GSK1437173A 50-70 Years Old Group
Number analyzed (Participants) | 3 | 20
gE-specific CD4 cells/million CD4 cells | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 3). | 899.8 (844.4)

4. Primary Outcome: Frequencies of Varicella Zoster Virus (VZV)-Specific CD4 / CD8 T Cells With at Least Two Antigen-specific Cytokines (IFN-γ, IL-2, TNF-α, CD40L).
Description: as for outcome 2
Time Frame: At Month 42 after the first vaccination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: VZV-specific CD4 cells/million CD4 cells
Arm/Group | GSK1437173A 18-30 Years Old Group | GSK1437173A 50-70 Years Old Group
Number analyzed (Participants) | 3 | 20
VZV-specific CD4 cells/million CD4 cells | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 3). | 723.8 (816.4)

5. Secondary Outcome: Frequencies of gE- and VZV-specific CD4/CD8 T Cells With Antigen-specific IFN-γ and/or IL-2 and/or TNF-α and/or CD40L Secretion/Expression.
Description: The analysis focused on those gE- and VZV-specific CD4 T cells secreting any cytokines among IFN-γ, IL-2, TNF-α, CD40L as determined by intracellular cytokine staining (ICS). No analysis of the immunogenicity data on CD8 T cell response to gE or VZV was performed, since no long-term vaccine effect on gE- and VZV-specific CD8 T cell response was detected.
Time Frame: At Months 30 and 42 after the first vaccination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CD4 cells/million T-cells
Arm/Group | GSK1437173A 18-30 Years Old Group | GSK1437173A 50-70 Years Old Group
Number analyzed (Participants) | 4 | 29
CD4 cells/million T-cells
  gE, IL-2 and IFN-γ/TNF-α/CD40L, Month 30 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 1144.8 (912.2)
  gE, IFN-γ and IL-2/TNF-α/CD40L, Month 30 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 574.2 (402.7)
  gE, TNF-α and IFN-γ/IL-2/CD40L, Month 30 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 806.4 (721.1)
  gE, CD40L and IFN-γ/IL-2/TNF-α, Month 30 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 1173.8 (918.6)
  gE, IL-2 and IFN-γ/TNF-α/CD40L, Month 42: number analyzed (Participants) | 3 | 20
  gE, IL-2 and IFN-γ/TNF-α/CD40L, Month 42 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 896.9 (822.9)
  gE, IFN-γ and IL-2/TNF-α/CD40L, Month 42: number analyzed (Participants) | 3 | 20
  gE, IFN-γ and IL-2/TNF-α/CD40L, Month 42 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 531.5 (533.3)
  gE, TNF-α and IFN-γ/IL-2/CD40L, Month 42: number analyzed (Participants) | 3 | 20
  gE, TNF-α and IFN-γ/IL-2/CD40L, Month 42 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 506.5 (550.8)
  gE, CD40L and IFN-γ/IL-2/TNF-α, Month 42: number analyzed (Participants) | 3 | 20
  gE, CD40L and IFN-γ/IL-2/TNF-α, Month 42 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 855.5 (769.7)
  VZV, IL-2 and IFN-γ/TNF-α/CD40L, Month 30 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 654.2 (494.0)
  VZV, IFN-γ and IL-2/TNF-α/CD40L, Month 30 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 467.1 (349.9)
  VZV, TNF-α and IFN-γ/IL-2/CD40L, Month 30 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 528.0 (417.3)
  VZV, CD40L and IFN-γ/IL-2/TNF-α, Month 30 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 694.2 (518.3)
  VZV, IL-2 and IFN-γ/TNF-α/CD40L, Month 42 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 631.5 (694.6)
  VZV, IFN-γ and IL-2/TNF-α/CD40L, Month 42 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 542.0 (682.1)
  VZV, TNF-α and IFN-γ/IL-2/CD40L, Month 42 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 556.1 (629.9)
  VZV, CD40L and IFN-γ/IL-2/TNF-α, Month 42 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 617.3 (743.6)

6. Secondary Outcome: Anti-gE Antibody (Ab) Concentrations
Description: As determined by the Enzyme-Linked Immunosorbent Assay (ELISA) and expressed as ELISA units per milliliter (EL.U/mL).
Time Frame: At months 30 and 42 after the first vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK1437173A 18-30 Years Old Group | GSK1437173A 50-70 Years Old Group
Number analyzed (Participants) | 4 | 29
EL.U/mL
  At Month 30 | 4008.9 [2048.0 to 7847.1] | 3390.1 [2684.9 to 4280.6]
  At Month 42: number analyzed (Participants) | 3 | 20
  At Month 42 | 3662.2 [905.6 to 14809.0] | 2413.1 [1698.8 to 3427.8]

7. Secondary Outcome: Anti-VZV Ab Concentrations
Description: As determined by the Enzyme-Linked Immunosorbent Assay (ELISA) and expressed as ELISA units per milliliter (EL.U/mL).
Time Frame: At months 30 and 42 after the first vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK1437173A 18-30 Years Old Group | GSK1437173A 50-70 Years Old Group
Number analyzed (Participants) | 4 | 29
EL.U/mL
  At Month 30 | 5341.8 [2247.8 to 12694.5] | 4049.3 [3340.0 to 4909.2]
  At Month 42: number analyzed (Participants) | 3 | 20
  At Month 42 | 3988.2 [753.2 to 21115.9] | 2683.3 [1991.2 to 3615.9]

8. Secondary Outcome: Frequencies of gE-specific Memory B Cells
Description: As determined by Enzyme-Linked ImmunoSpot (ELISPOT) assay.
Time Frame: At months 30 and 42 after the first vaccination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gE-specific B-cells/million B-cells
Arm/Group | GSK1437173A 18-30 Years Old Group | GSK1437173A 50-70 Years Old Group
Number analyzed (Participants) | 4 | 29
gE-specific B-cells/million B-cells
  At Month 30: number analyzed (Participants) | 4 | 27
  At Month 30 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 3614.2 (2389.8)
  At Month 42: number analyzed (Participants) | 3 | 20
  At Month 42 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 2696.1 (2644.0)

9. Secondary Outcome: Frequencies of VZV-specific Memory B Cells
Description: As determined by Enzyme-Linked ImmunoSpot (ELISPOT) assay.
Time Frame: At months 30 and 42 after the first vaccination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: VZV-specific B-cells/million B-cells
Arm/Group | GSK1437173A 18-30 Years Old Group | GSK1437173A 50-70 Years Old Group
Number analyzed (Participants) | 4 | 29
VZV-specific B-cells/million B-cells
  At Month 30: number analyzed (Participants) | 4 | 27
  At Month 30 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 4853.8 (3362.1)
  At Month 42: number analyzed (Participants) | 3 | 20
  At Month 42 | NA (NA) — Descriptive statistics on immune persistence data in the GSK1437173A 18-30 Years Old Group were not performed, since the number of enrolled subjects in this age cohort was too low (N = 4 at M30 and N = 3 at M42). | 3488.1 (2689.1)

10. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of existing hospitalization, result in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Month 30 to study end Month 42 after the first vaccination
Population: The analysis was performed on the Total cohort for persistence which included all subjects previously primed with 2 doses of GSK1437173A and were enrolled in the current study.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A 18-30 Years Old Group | GSK1437173A 50-70 Years Old Group
Number analyzed (Participants) | 4 | 30
Participants | 0 | 0

11. Secondary Outcome: Number of Subjects With Clinically Diagnosed Herpes Zoster (HZ) Episodes
Description: This assay tabulated the number of subjects with clinically diagnosed HZ episodes, defined as any cutaneous HZ-like rash.
Time Frame: From last primary study visit (Month 12) to study end at Month 42 after the first vaccination.
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A 18-30 Years Old Group | GSK1437173A 50-70 Years Old Group
Number analyzed (Participants) | 4 | 30
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected throughout the study, up to Month 42.
Description: Other (Not Including Serious) Adverse Events were not planned to be collected in this study.
Arm/Group | GSK1437173A 18-30 Years Old Group | GSK1437173A 50-70 Years Old Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/30
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.